CLINICAL TRIAL: NCT05123638
Title: Is Virtual Reality Assisted Cycling Exercise Superior to Conventional Stationary Cycling in Geriatric Patients for Increasing Physical Activity Levels During Hospitalization?
Brief Title: VR vs. Conventional Cycling Exercise for Geriatric Inpatient Physical Activation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Suetta, Clinical professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VR+Cycling
Record Dates: First submitted 2021-11-06; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Inactivity, Physical; Treatment Adherence and Compliance; Hospital Acquired Condition; Sarcopenia
Keywords: Virtual Reality; Patient Preference
MeSH Terms: conditions — Sedentary Behavior; Treatment Adherence and Compliance; Iatrogenic Disease; Sarcopenia; Patient Preference

STUDY DESIGN:
Intervention Model Description: Stratified randomization (based os Cumulated-Ambulation Score of 6 vs. <6) of geriatric inpatients to either VR assisted stationary cycling exercise or conventional stationary cycling exercise.
Masking Description: Since there is only a single investigator conducting this study and due to the nature of exercise intervention, it is impossible to facilitate masking terms in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality cycling exercise (Experimental): These patient participants will receive 1 session of unsupervised stationary cycling exercise with the SYNCSENSE VR-technology every weekday of participation and be allowed up to 30min of voluntary exercise pr. session.
  Interventions: Device: Virtual reality cycling exercise
- Conventional cycling exercise (Active Comparator): These patient participants will receive 1 session of unsupervised stationary cycling exercise on every weekday of participation and be allowed up to 30min of voluntary exercise pr. session.
  Interventions: Behavioral: Unsupervised stationary cycling exercise

INTERVENTIONS:
Device: Virtual reality cycling exercise — Daily voluntary cycling for up to 30 minutes with the virtual reality technology
  Arms: Virtual reality cycling exercise
Behavioral: Unsupervised stationary cycling exercise — Daily voluntary cycling for up to 30 minutes (WITHOUT the virtual reality technology)
  Arms: Conventional cycling exercise

SUMMARY:
The aim of this study is to investigate whether virtual reality assisted stationary cycling exercise results in more physical activity than conventional unsupervised stationary cycling exercise. Physical activity levels are reported for both exercise duration and volume and non-exercise activity.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to geriatric ward at Bispebjerg Hospital with an minimum of 3 days (anticipated) left of stay.
* Volunteering

Exclusion Criteria:

* Unable to be easily mobilized by training staff.
* Unable to perform the stationary cycling exercise modality.
* Lack of Danish speaking and reading skills.
* Lack of senses (blind, deff pr heavily hearing impaired).
* Suffering from delirium, vertigo or dementia beyond a moderate degree.
* Judged medically contraindicated by therapeutic, medical or care staff

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-08 (Estimated); Primary Completion 2021-12-22 (Estimated); Study Completion 2022-01-07 (Estimated)

PRIMARY OUTCOMES:
Voluntary exercise duration | 3-14 days
  How long the patients choose to exercise with vs. with out VR assistance measured on the stationary bikes internal timer

SECONDARY OUTCOMES:
Voluntary exercise amount | 3-14 days
  How much voluntary cycling work does the participants choose to put out during session calculated from the bikes internal counter and external equations
Measures of 24 hour physical activity and sedentary behavior | 3-14 days
  Measured with 24 hour thigh mounted movement sensor

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suetta, Study Director — CopenAge
Locations (1):
- Bispebjerg Geriatric Ward, Bispebjerg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
It is wanted but not yet premised